CLINICAL TRIAL: NCT03375216
Title: Quantitative Sensory Testing in Chronic Pain Patients Undergoing Opioid Treatment and Opioid Tapering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0195
Record Dates: First submitted 2017-12-05; First posted 2017-12-15 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Analgesic Drug Dependence; Sensory Deficit
MeSH Terms: interventions — Hot Temperature; Cold Temperature; Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- taper (Active Comparator): participants undergoing a taper as directed by their pain physician. Interventions include sensory testing ( heat, cold, and pressure) and PROMIS surveys.
  Interventions: Behavioral: sensory testing (Heat, cold, and pressure); Behavioral: Promis Survey
- non taper systemic <90 (Placebo Comparator): participants on systemic opioids < 90 MEDD (morphine equivalent daily dose) and no taper
  Interventions: Behavioral: sensory testing (Heat, cold, and pressure); Behavioral: Promis Survey
- non taper systemic >90 (Placebo Comparator): participants on systemic opioids > 90 MEDD and no taper
  Interventions: Behavioral: sensory testing (Heat, cold, and pressure); Behavioral: Promis Survey
- non taper intrathecal (Placebo Comparator): Participants on intrathecal therapy and no taper
  Interventions: Behavioral: sensory testing (Heat, cold, and pressure); Behavioral: Promis Survey
- non opioids (Sham Comparator): Participants on non-opioid therapy will undergo behavioral tests and PROMIS surveys
  Interventions: Behavioral: sensory testing (Heat, cold, and pressure); Behavioral: Promis Survey

INTERVENTIONS:
Behavioral: sensory testing (Heat, cold, and pressure) — sensory threshold measurement is the point at which the participant feels pain due to either heat, cold, or pressure
Behavioral: Promis Survey — PROMIS computer adaptive survey in anxiety, depression, pain behavior, fatigue, pian interference, physical function, sleep disturbance, self efficacy

SUMMARY:
Few studies have used quantitative sensory tests to study the effect of chronic opioid treatment on sensation. The investigators will test chronic pain patients who are on different MEDDs, normal volunteers, and patients undergoing an opioid taper. This will be the first study to perform sensory testing on patients while undergoing an opioid taper on an outpatient basis.

DETAILED DESCRIPTION:
Death from drug overdoses reached a record high in 2014, with the majority involving an opioid. The United States government has labeled this an epidemic due to the progressive rise in opioid-involved deaths. In 2015, the Centers for Disease Control and Prevention determined that, on average, 650,000 opioid prescriptions are dispensed daily in the United States alone. It is well-documented and observed in clinical practice that patients on chronic opioid therapy will commonly require an escalation in opioid dose over time to maintain analgesia. The consequence of such escalations is the development of tolerance to opioids, along with other known adverse effects of opioids including respiratory depression, constipation, and potential for addiction. The drastic increase in opioid doses over the years has urged the CDC to release a report for primary care clinicians treating patients with chronic pain. This report provides a risk assessment and recommendations for prescribing opioids for non-cancer chronic pain. The guidelines state that careful reassessment of individual benefits must be considered when increasing doses to ≥50 morphine milligram equivalents (MME)/day, and that increases to ≥90 MME/day must be avoided, with recommendations for consultation with a specialist. Avoiding high opioid doses will also minimize the development of opioid-induced hyperalgesia, which is a paradoxical response to increases in opioid doses; these patients become increasingly sensitized to painful stimuli. While the precise mechanism of this condition remains to be elucidated, treatment includes reducing and tapering opioids. Interestingly, an article on patient-reported outcomes surveyed a group of 517 patients that revealed the higher opioid dose group to have greater pain intensity, poorer self-efficacy for managing pain, and more impairment in functioning and quality of life.

Several studies have looked at the use of various pain testing models to investigate the effects of chronic opioid therapy and changes in pain perception. A systematic review of the literature was performed to identify clinical studies incorporating measures of hyperalgesia in patients on chronic opioid therapy. This review was aimed at finding the optimal testing modality to evaluate pain threshold and tolerance to external stimuli, including mechanical (pressure, touch, injection), thermal (cold/heat), and electrical. Although the results did not reveal any one method with sufficient power, several prospective studies evaluating hyperalgesia with heat pain ratings have shown some promising results; two studies revealing significant changes in heat responses for opioid treatment groups, and one study demonstrating lower heat pain perception values following an opioid taper. The latter study is unique in that research pertaining to changes in pain sensitivity on patients following an opioid taper is lacking. Little is known at this juncture how pain thresholds change to opioid dose reductions and following completion of a taper.

The purpose of the study is to objectively measure pain threshold levels in patients without opioids, low dose opioids, high dose opioids and patients undergoing a taper from long-term opioid therapy. This study utilizes taper techniques that are commonly employed in a pain medicine practice. The innovation involves use of quantitative measures of sensitivity to evaluate patients on differing opioid doses and undergoing current taper practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 18 and 75
* History of chronic pain for at least 3 months
* Patients may have been selected for opioid taper by their pain physicians.
* Patients may or may not be on opioid therapy.
* They must have the ability to understand the protocol and provide voluntary, written, informed consent.

Exclusion Criteria:

* Cancer pain
* Unstable medical conditions (including but not limited to history of myocardial infarction within the past year, autoimmune diseases, uncontrolled diabetes with hemoglobin A1C of greater than 10)
* Pregnancy
* Inability to adequately answer surveys
* History of substance abuse within 5 years
* Surgery within the past month
* Surgery planned during the next six months
* Use of systemic steroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Heat threshold measurements | 2 years
  Heat threshold measurements (degrees Celsius) will be obtained using a pen-shaped temperature probe. Tests will be performed on a designated painful and non-painful body surface. Testing will completed when patient reports numeric pain rating of 5 or greater, or at a temperature >49 degrees Celsius.
Cold threshold measurements | 2 years
  Cold threshold measurements (degrees Celsius) will be obtained using a pen-shaped temperature probe. Tests will be performed on a designated painful and non-painful body surface. Testing will be completed when patient reports discomfort with cold stimulus, or if probe temperature reaches 0 degrees Celsius.
Pressure threshold measurements | 2 years
  Pressure threshold measurements (Newtons) will be obtained using a hand-held algometer. Tests will be performed on a designated painful and non-painful body surface. Testing will be completed when patient reports discomfort with pressure stimulus, or if pressure exceeds 60 Newtons.

SECONDARY OUTCOMES:
PROMIS surveys | 2 years
  PROMIS (Patient-Reported Outcomes Measurement Information System) surveys will be administered at the subject's initial, halfway and end of their evaluations. These measures include topics on anxiety, depression, pain behavior, fatigue, pain interference, physical function, sleep disturbance. The results from the surveys will be aggregated and compared to other participants' responses.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilkes, MD-PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Result] Chu LF, D'Arcy N, Brady C, Zamora AK, Young CA, Kim JE, Clemenson AM, Angst MS, Clark DJ. Analgesic tolerance without demonstrable opioid-induced hyperalgesia: a double-blinded, randomized, placebo-controlled trial of sustained-release morphine for treatment of chronic nonradicular low-back pain. Pain. 2012 Aug;153(8):1583-1592. doi: 10.1016/j.pain.2012.02.028. Epub 2012 Jun 16. PMID 22704854
- [Result] Dumas EO, Pollack GM. Opioid tolerance development: a pharmacokinetic/pharmacodynamic perspective. AAPS J. 2008 Dec;10(4):537-51. doi: 10.1208/s12248-008-9056-1. Epub 2008 Nov 7. PMID 18989788
- [Result] Dyck PJ, Zimmerman IR, Johnson DM, Gillen D, Hokanson JL, Karnes JL, Gruener G, O'Brien PC. A standard test of heat-pain responses using CASE IV. J Neurol Sci. 1996 Mar;136(1-2):54-63. doi: 10.1016/0022-510x(95)00277-9. PMID 8815179
- [Result] Hooten WM, Mantilla CB, Sandroni P, Townsend CO. Associations between heat pain perception and opioid dose among patients with chronic pain undergoing opioid tapering. Pain Med. 2010 Nov;11(11):1587-98. doi: 10.1111/j.1526-4637.2010.00962.x. Epub 2010 Oct 1. PMID 21029354
- [Result] Katz NP, Paillard FC, Edwards RR. Review of the performance of quantitative sensory testing methods to detect hyperalgesia in chronic pain patients on long-term opioids. Anesthesiology. 2015 Mar;122(3):677-85. doi: 10.1097/ALN.0000000000000530. PMID 25437498
- [Result] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Result] Morasco BJ, Yarborough BJ, Smith NX, Dobscha SK, Deyo RA, Perrin NA, Green CA. Higher Prescription Opioid Dose is Associated With Worse Patient-Reported Pain Outcomes and More Health Care Utilization. J Pain. 2017 Apr;18(4):437-445. doi: 10.1016/j.jpain.2016.12.004. Epub 2016 Dec 18. PMID 27993558
- [Result] Pud D, Cohen D, Lawental E, Eisenberg E. Opioids and abnormal pain perception: New evidence from a study of chronic opioid addicts and healthy subjects. Drug Alcohol Depend. 2006 May 20;82(3):218-23. doi: 10.1016/j.drugalcdep.2005.09.007. Epub 2005 Oct 17. PMID 16229972
- [Result] Krishnan S, Salter A, Sullivan T, Gentgall M, White J, Rolan P. Comparison of pain models to detect opioid-induced hyperalgesia. J Pain Res. 2012;5:99-106. doi: 10.2147/JPR.S27738. Epub 2012 Apr 27. PMID 22570562
- [Result] Sullivan MD, Turner JA, DiLodovico C, D'Appollonio A, Stephens K, Chan YF. Prescription Opioid Taper Support for Outpatients With Chronic Pain: A Randomized Controlled Trial. J Pain. 2017 Mar;18(3):308-318. doi: 10.1016/j.jpain.2016.11.003. Epub 2016 Nov 28. PMID 27908840
- [Result] Suzan E, Eisenberg E, Treister R, Haddad M, Pud D. A negative correlation between hyperalgesia and analgesia in patients with chronic radicular pain: is hydromorphone therapy a double-edged sword? Pain Physician. 2013 Jan;16(1):65-76. PMID 23340535
- [Result] Wasserman RA, Hassett AL, Harte SE, Goesling J, Malinoff HL, Berland DW, Zollars J, Moser SE, Brummett CM. Pressure Pain Sensitivity in Patients With Suspected Opioid-Induced Hyperalgesia. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):687-93. doi: 10.1097/AAP.0000000000000315. PMID 26469365
- [Result] Weimer MB, Hartung DM, Ahmed S, Nicolaidis C. A chronic opioid therapy dose reduction policy in primary care. Subst Abus. 2016;37(1):141-7. doi: 10.1080/08897077.2015.1129526. PMID 26685018
- [Result] Wilkes D, Martinello C, Medeiros FA, Babazade R, Hurwitz E, Khanjee N, Iyer PS, Leary P, Vadhera RB. Ultrasound-determined landmarks decrease pressure pain at epidural insertion site in immediate post-partum period. Minerva Anestesiol. 2017 Oct;83(10):1034-1041. doi: 10.23736/S0375-9393.17.11782-7. Epub 2017 Apr 11. PMID 28402092
- [Result] Wright A, Benson HAE, Will R, Moss P. Cold Pain Threshold Identifies a Subgroup of Individuals With Knee Osteoarthritis That Present With Multimodality Hyperalgesia and Elevated Pain Levels. Clin J Pain. 2017 Sep;33(9):793-803. doi: 10.1097/AJP.0000000000000458. PMID 27898461
- See also: MMWR Recomm Rep 2016 — http://dx.doi.org/10.15585/mmwr.rr6501e1